CLINICAL TRIAL: NCT06832215
Title: Urine Extracellular Vesicles: Non-invasive Biomarkers of Β-cell Function and Novel Therapeutic Agents in Diabetes
Acronym: EvsBioDiabetes
Status: Active, not recruiting | Type: Observational
Sponsor: Unidade Local de Saúde de Coimbra, EPE (Other)
Collaborators: Università di Siena (Unknown)
Responsible Party: Principal Investigator, Joana Serra Caetano, MD, Consultant in Pediatrics (Graduated), Pediatric Endocrinologist and Diabetologist, Unidade Local de Saúde de Coimbra, EPE
Other Study IDs: OBS.SF.05.2023
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus
Keywords: Non-invasive biomarker of beta cell function in urine
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Type 1 Diabetes Group: Type 1 Diabetes people under 18 years´old
  Interventions: Diagnostic Test: Blood and urine samples collection
- Genetic-related Group: Brothers/sisters of T1D children and adolescents (without disease)
  Interventions: Diagnostic Test: Blood and urine samples collection
- Control group: Not genetic related and no T1D people under 18 years' old
  Interventions: Diagnostic Test: Blood and urine samples collection

INTERVENTIONS:
Diagnostic Test: Blood and urine samples collection — Blood and urine were collected at a single time point for all participants, from the tree study groups. Fasting for blood collection and the first urine in the morning were required.

SUMMARY:
Diabetes mellitus is a common chronic disease with a huge socioeconomic burden worldwide. Type 1 Diabetes(T1D) accounts for nearly 95% of diabetes in pediatric age and a lifelong dependence on exogenous insulin. Its diagnosis is based on symptoms and/or autoantibodies, both identified too late to avoid the disease progress. Ideally, children should be screened whilst assymptomatic, when there is endogenous insulin production, but C-peptide and beta-cell function are starting to decline. Early diagnosis would allow interventions capable of preventing disease progress and/or to preserve beta-cell function, ultimately delaying/avoiding insulin dependence. Given their association with pathogenesis of diabetes, Extracellular Vesicles have emerged as potential biomarkers for diagnosis and progression of diabetes. This project proposes the development of a non-invasive biomarker of preclinical T1D, based on miRNA characterization in urine, allowing a timely identification of children that can benefit from preventive therapies and, in the future, to cure T1D.

ELIGIBILITY:
Inclusion Criteria:

* T1D Group: children diagnosed with T1D, according to internationally defined criteria, with at least one positive pancreatic antibody and under functional insulin.
* Genetic-related group: children without T1D, age- and sex-matched with T1D group, recruited among T1D relatives;
* Control group: children without T1D, age- and sex-matched with T1D group, recruited from general endocrinology clinics, among children without disease or genetic relation with T1D children;

Exclusion Criteria:

* Obesity, according to WHO standards for pediatrics;
* Hypertension, as ≥95th percentile according to International Consensus;
* Other auto-immune diseases;
* Diabetes in the context of syndromic features/secondary to treatments;
* Hypothyroidism, adrenal insufficiency or hypercortisolism;
* Children under somatotropin/oncologic treatment;
* Under medications affecting glucose metabolism

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children and adolescents under follow-up at Coimbra Pediatric Hospital - Coimbra University and Hospital Centre (CHUC), either in specific clinic (Diabetes - for T1D group) or that have been observed at a general endocrine or pediatrics clinics for a suspition of disease that was not confirmed (for control group). For the genetic related group, children and adolescents were recruited within T1D families and were observed in a single time point, at the time of their brother/sister.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-05-06 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Urine miRNAs extracellular vesicles molecular signatures for the study groups | October/23 until July/2024
  Characterize urine EV-derived miRNAs in the three study groups
Blood miRNAs extracellular vesicles molecular signatures for the study groups | October/23 until July/2024
  Characterize blood miRNAs extracellular vesicles molecular signatures for the study groups

CONTACTS AND LOCATIONS:
Locations (1):
- Coimbra Pediatric Hospital - CHUC, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No
Confidential information collected with permission for this study purpose but not to share with other studies